CLINICAL TRIAL: NCT02434198
Title: Falling in Patients With COPD Referred to Pulmonary Rehabilitation: Incidence, Risk Factors and Prediction Tools
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Thierry Troosters, Prof, KU Leuven
Other Study IDs: S57678
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: pulmonary rehabilitation; balance assessment; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim of this study is to investigate the incidence of falling in a cohort of patients with chronic obstructive pulmonary disease (COPD) referred to a pulmonary rehabilitation program and to verify the risk factors. The secondary aim is to verify whether available balance assessment tools are feasible in clinical practice and which tools and values can best predict falls in people with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of COPD according to internationally accepted guidelines
* All patients referred to the outpatient PR program of Gasthuisberg University Hospital (Leuven, Belgium).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred to the outpatient pulmonary rehabilitation (PR) program in the Gasthuisberg University Hospital (Leuven, Belgium) will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
incidence of falling | 6 months

SECONDARY OUTCOMES:
association between falling status and the score in balance tests | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Troosters, PhD, Principal Investigator — KU Leuven
Locations (1):
- University hospitals Leuven, Leuven, Vlaams Brabant, Belgium